CLINICAL TRIAL: NCT03035565
Title: Cognitive Intervention to Improve Memory in Heart Failure Patients
Acronym: Memoir-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Susan Pressler, Principal Investigator, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR016116-01A1 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-30 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class I
Keywords: Heart Failure; Cognition in Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computerized Cognitive Training Brain HQ (Experimental): Computerized cognitive training intervention using Brain HQ initiated and continued 1 hour/day, 5 days/week for 8 weeks
  Interventions: Behavioral: Computerized Cognitive Training with Brain HQ
- Computerized Crossword Puzzles (Active Comparator): General cognitive stimulation puzzles intervention initiated and continued 1 hour/day, 5 days/week for 8 weeks
  Interventions: Behavioral: Computerized Crossword Puzzles
- Usual Care (No Intervention): No computerized cognitive intervention

INTERVENTIONS:
Behavioral: Computerized Cognitive Training with Brain HQ — Computerized Cognitive Training Brain HQ activities initiated and continued 1 hour/day, 5 days/week for 8 weeks
  Arms: Computerized Cognitive Training Brain HQ
Behavioral: Computerized Crossword Puzzles — Computerized Crossword Puzzles activities initiated and continued 1 hour/day, 5 days/week for 8 weeks
  Arms: Computerized Crossword Puzzles

SUMMARY:
Cognitive Intervention to Improve Memory in Heart Failure patients

DETAILED DESCRIPTION:
A three arm randomized controlled trial of 276 heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Understands English
* Has access to a telephone
* Hears normal conversation
* For patients with hearing aids, able to wear and hear through headsets
* Diagnosis of chronic heart failure, stage C, NYHA I, II or III
* Receiving guideline derived medical therapy
* Heart failure validated by echocardiography or other method in past 2 years
* Able to read a computer screen with or without glasses or lenses

Exclusion Criteria:

* History of drug or alcohol abuse or major psychiatric diagnosis present before the heart failure diagnosis
* Alzheimer or other dementia diagnosis or central nervous system degenerative disorder
* Terminal cancer
* Patients with baseline Montreal Cognitive Assessment (MoCA) score of less than 19

Supplement Eligibility: First 144 patients randomized in the parent trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in delayed recall memory as measured by Hopkins Verbal Learning Test | At 8 months
  Change in delayed recall memory as measured by Hopkins Verbal Learning Test
Change in serum brain derived neurotrophic factor ( BDNF) Level | At 8 months
  Co-Primary Outcome

SECONDARY OUTCOMES:
Change in working memory as measured by CogState One Back Accuracy Task | At 8 months
  Change in working memory as measured by CogState One Back Accuracy Task
Change in instrumental activities of daily living as measured by Everyday Problems Test | At 8 months
  Change in instrumental activities of daily living as measured by Everyday Problems Test
Change in health-related quality of life as measured by Minnesota Living with Heart Failure Questionnaire | At 8 months
  Change in health-related quality of life as measured by Minnesota Living with Heart Failure Questionnaire
Cost-effectiveness of the Brain HQ training intervention as measured by calculating the Incremental cost effectiveness ratios (ICERs) using medical services costs | At 8 months
  Cost-effectiveness of the Brain HQ training intervention as measured by calculating the Incremental cost effectiveness ratios (ICERs) using medical services costs

OTHER OUTCOMES:
Cognitive Intervention to Improve Memory in Heart Failure Patients - Supplement | Across 36 months
  Risk of amnestic mild cognitive impairment, Alzheimer disease and related dementias, and memory decline across 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Pressler, PhD, RN, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Health, Indianapolis, Indiana
  - Methodist Hospital-Krannert Institute of Cardiology, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Pressler SJ, Giordani B, Titler M, Gradus-Pizlo I, Smith D, Dorsey SG, Gao S, Jung M. Design and Rationale of the Cognitive Intervention to Improve Memory in Heart Failure Patients Study. J Cardiovasc Nurs. 2018 Jul/Aug;33(4):344-355. doi: 10.1097/JCN.0000000000000463. PMID 29601367
- [Background] Algashgari EY, Jung M, Von Ah D, Stewart JC, Pressler SJ. Perceived Facilitators and Barriers to Treatment Fidelity in Computerized Cognitive Training Interventions. J Cardiovasc Nurs. 2022 Apr 20. doi: 10.1097/JCN.0000000000000916. Online ahead of print. PMID 35467571
- [Background] Halloway S, Jung M, Yeh AY, Liu J, McAdams E, Barley M, Dorsey SG, Pressler SJ. An Integrative Review of Brain-Derived Neurotrophic Factor and Serious Cardiovascular Conditions. Nurs Res. 2020 Sep/Oct;69(5):376-390. doi: 10.1097/NNR.0000000000000454. PMID 32555009
- [Result] Pressler SJ, Jung M, Gradus-Pizlo I, Titler MG, Smith DG, Gao S, Lake KR, Burney H, Clark DG, Wierenga KL, Dorsey SG, Giordani B. Randomized Controlled Trial of a Cognitive Intervention to Improve Memory in Heart Failure. J Card Fail. 2022 Apr;28(4):519-530. doi: 10.1016/j.cardfail.2021.10.008. Epub 2021 Nov 8. PMID 34763080
- [Derived] Smith AB, Jung M, Pressler SJ, Mocci E, Dorsey SG. Differential Gene Expression Among Patients With Heart Failure Experiencing Pain. Nurs Res. 2023 May-Jun 01;72(3):175-184. doi: 10.1097/NNR.0000000000000648. Epub 2023 Feb 26. PMID 36920122